CLINICAL TRIAL: NCT01637337
Title: Laparoscopic Pyelolithotomy Versus Percutaneous Nephrolothotomy for Management of >3cm Renal Pelvis Stone
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Aminsharifi, Assistant Professor of Urology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 89-01-01-2391
Record Dates: First submitted 2012-07-03; First posted 2012-07-11 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Renal Pelvis Stone >3cm
MeSH Terms: interventions — Nephrolithotomy, Percutaneous

ARMS (2):
- laparoscopic pyelolithotomy (Active Comparator)
  Interventions: Procedure: laparoscopic pyelolithotomy
- percutaneous nephrolithotomy (Sham Comparator)
  Interventions: Procedure: percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: laparoscopic pyelolithotomy — laparoscopy
  Arms: laparoscopic pyelolithotomy
Procedure: percutaneous nephrolithotomy — percutaneous nephrolithotomy
  Arms: percutaneous nephrolithotomy

SUMMARY:
To compare the outcome of laparoscopic pyelolithotomy with percutaneous nephrolithotomy in patients with >3cm renal pelvis stone.

ELIGIBILITY:
Inclusion Criteria:

* Adults with >3cm renal pelvis stone

Exclusion Criteria:

* History of previous surgery on the target kidney
* Active UTI
* Coagulopathy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Stone free rate | at least 6 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran